CLINICAL TRIAL: NCT04078048
Title: Role of Selected Antioxidants (Vitamin C and E) in the Management of Schizophrenia
Brief Title: Role of Antioxidants (Vitamin C and E) in the Management of Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Saima Zahid, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: UHS
Record Dates: First submitted 2019-09-01; First posted 2019-09-04 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia
Keywords: Positive and Negative syndrome scale (PANSS); Antioxidants; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Antioxidants; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vitamin C Group (Experimental): Tablet Vitamin C 500 mg Once a day
  Interventions: Dietary Supplement: Antioxidants (Vitamin C, E )
- Vitamin E Group (Experimental): Tablet Vitamin E 600 I U Twice daily
  Interventions: Dietary Supplement: Antioxidants (Vitamin C, E )
- Placebo Group (Placebo Comparator): Capsule Paraffin oil 500 mg Once a day
  Interventions: Dietary Supplement: Antioxidants (Vitamin C, E )

INTERVENTIONS:
Dietary Supplement: Antioxidants (Vitamin C, E ) — For eight weeks, Vitamin C group was intervened with tablet vitamin c 500 mg once a day ,vitamin E group was intervened with Tablet vitamin E 600 I U twice a day.
  Other Names: Tablet Vitamin E

SUMMARY:
Background: Antioxidants are substances that are considered as a defensive material which protects cells from destruction. It is evident that use of food stuff rich in antioxidant will fortify one's ability to encounter with physical & mental disorders. Since, among several potential elucidations, oxidative stress is more likely deliberated as one of the causative factors which give rise to cognitive and functional impairment. This deterioration further result in intricacy in ones thought process as progressive brain changes crop-up schizophrenic unfold. Therefore, this study was conducted with objectives to explore the role of selected antioxidants (vitamin C & E) and to compare the role of both vitamins as an add-on management of schizophrenia .Materials & Methods: One hundred and five patients were selected from department of psychiatry King Edward Medical University Lahore, and assigned into 3 groups by simple random lottery method. For eight weeks, Vitamin C group intervened with 500mg vitamin C tablet once a day, vitamin E group with 600IU vitamin E twice daily and placebo group was given 500 mg paraffin oil capsule daily. PANSS scale was used to assess the symptoms of schizophrenia. Demographic information was collected by structured questionnaire. Dietary habits were assessed by food frequency questionnaire.

DETAILED DESCRIPTION:
Background: Antioxidants such as Vitamin C and E are substances that are considered as a defensive material which protects cells from destruction. It is evident that use of food stuff rich in antioxidant will fortify one's ability to encounter with physical & mental disorders. Since, among several potential elucidations, oxidation stress is more likely deliberated as one of the causative factors which give rise to cognitive and functional impairment. Therefore, this study was conducted with objectives to explore the role of selected antioxidants (vitamin C & E) and to compare the role of both vitamins as an add-on management of schizophrenia .Materials & Methods: One hundred and five patients were selected from department of psychiatry King Edward Medical University Lahore, and assigned into 3 groups by simple random lottery method. For the period of two months, Vitamin C group intervened with 500 mg vitamin C tablet once a day, vitamin E group with 600 I U vitamin E twice daily and placebo group was given 500 mg paraffin oil capsule daily. PANSS (Positive and Negative Symptoms Scale) was used to assess the symptoms of schizophrenia. Demographic information was collected by structured questionnaire. Dietary habits were assessed by (FFQ) food frequency questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA:

  * All diagnosed schizophrenic patients 20-50 years of age
  * visited department of psychiatry & behavioral sciences King Edward medical university Lahore.
* EXCLUSION CRITERIA:

  * Patients diagnosed with axis i and axis ii disorders
  * having any other pathological condition like hypertension, hyperlipidemia, and cardiac disorders.

Exclusion Criteria:

-

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale | 45-50 minutes
  The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of patients with schizophrenia.The PANSS yields a total average symptom score, based on 30 items rated from one to seven (range=30-210). Higher scores indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Saima Kouser, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
clinical trails registration